CLINICAL TRIAL: NCT06969118
Title: A Multi-center, Randomized, Controlled Study Comparing Minimalist Procedure With Standard Procedure for Left Atrial Appendage Closure in Patients With Non-valvular Atrial Fibrillation
Brief Title: RCT of Minimalist vs Standard Procedure for LAAC in NVAF Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MVS-LAAC
Record Dates: First submitted 2024-08-30; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation; Left Atrial Appendage Occlusion; General Anesthesia; Local Anesthesia
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Minimalism Transcatheter LAAC Group (Experimental): Patients underwent LAAC under simplified guidance of TTE and fluoroscopy.
  Interventions: Procedure: Minimalism Transcatheter LAAC Group
- Standard Transcatheter LAAC Group (Placebo Comparator): Patients underwent LAAC under standard guidance of TEE and fluoroscopy.
  Interventions: Procedure: Standard Transcatheter LAAC Group

INTERVENTIONS:
Procedure: Minimalism Transcatheter LAAC Group — Patients will undergo transcatheter LAAC under local anesthesia, guided by DSA and TTE, using the WATCHMAN FLX system. The release criteria (PASS: Position, Anchor, Size, Seal) will be confirmed through DSA and TTE.
  Arms: Minimalism Transcatheter LAAC Group
Procedure: Standard Transcatheter LAAC Group — Patients will undergo LAAC under general anesthesia, guided by TEE, using the WATCHMAN FLX system, following the steps outlined in the product manual.
  Arms: Standard Transcatheter LAAC Group

SUMMARY:
Percutaneous left atrial appendage closure (LAAC) is an effective strategy for stroke prevention in patients with non-valvular atrial fibrillation (NVAF). Standard procedure requires general anesthesia, transesophageal echocardiography (TEE) guidance. With the experience accumulation, LAAC can be successfully completed in many centers under local anesthesia, the guidance of X-ray and transthoracic echocardiography (TTE), also known as minimalist procedure. Our center was one of the earliest to carry out minimalist procedure worldwide. At present, expert consensus suggests that minimalist procedure is feasible in experienced centers, but the relevant evidence is insufficient. Some single-arm studies have shown that minimalist procedure is safe and effective. However, there is currently a lack of direct evidence to compare the strengths and weaknesses of these two LAAC procedures. The goal of the study was to compare the effectiveness and safety of minimalist procedure and standard procedure for LAAC in patients with NVAF.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled, multi-center clinical study designed to compare the safety and efficacy of minimalism transcatheter LAAC versus standard transcatheter LAAC in NVAF patients. The study aims to enroll approximately 200 NVAF patients requiring transcatheter LAAC at 20 to 30 research centers in China. All eligible patients who sign the informed consent form will be randomly assigned to either the minimalism transcatheter LAAC group or the standard transcatheter LAAC group in a 1:1 ratio. The study will record preoperative baseline information and follow-up data at 7 days post-Procedure or discharge, and at 2, 6, and 12 months post-Procedure, to explore the incidence of procedure-related complications and peridevice leak ≤5mm between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 85 years old, all genders;
2. Subjects who can understand the purpose of the trial, participate voluntarily and sign the informed consent form, and are willing to complete the follow-up according to the protocol requirements;
3. Indications for left atrial appendage closure: non-valvular atrial fibrillation patients with CHA2DS2-VAS2 score ≥2 and HAS-BLED score ≥3, or who are unable or unwilling to receive long-term oral anticoagulants;
4. Life expectancy ≥1 year;

Exclusion Criteria:

1. Preoperative TEE/heart CT/intracardiac ultrasound suggested thrombus in the left atrial appendage/left atrium;
2. Patients with severe renal insufficiency (creatinine ≥200 μmol/L, creatinine clearance <30 ml/min);
3. Liver disease patients with coagulation abnormalities and clinically relevant bleeding risks, including liver cirrhosis patients reaching Child Pugh stages B and C;
4. Severely decreased platelet count at baseline: PLT ≤50*10^9/L;
5. Patients with severe preoperative cardiac insufficiency (LVEF <35%; clinical manifestations are uncontrolled class IV heart failure);
6. Combined with other severe cardiac valvular diseases or other structural abnormalities that require surgical treatment on an elective day; or severe coronary heart disease that requires intervention within a fixed period;
7. Patients who have lesions or conditions with a significant risk of major bleeding, such as current or recent gastrointestinal ulcers, malignant tumors with a high risk of bleeding, recent brain or spinal injuries, recent brain, spinal or ophthalmic procedure, recent intracranial hemorrhage, known or suspected esophageal varices, arteriovenous malformations, vascular aneurysms, or major intraspinal or intracerebral vascular malformations;
8. Patients with concurrent diseases (other than atrial fibrillation) that require anticoagulant therapy (such as after mechanical valve replacement, and spontaneous or recurrent venous thromboembolism);
9. Patients who are in clinical trials of other drugs or medical devices and have not completed it yet;
10. Patients who are considered ineligible to participate in the clinical trial by the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
primary safety | 7 days after LAAC procedure
  Occurrence of a composite endpoint about serious perioperative complications including all-cause death, ischemic or hemorrhagic stroke, systemic embolism, and procedure related complications requiring thoracotomy or endovascular intervention treatment.
primary efficacy | From LAAC procedure to the end of treatment at 12 months
  Occurrence of successful device implantation under predetermined guidance as well as effective LAA closure with residual leak ≤ 5mm

SECONDARY OUTCOMES:
Stroke/transient ischemic attack and systemic embolism | at 2, 6, and 12 months post-procedure
  Occurrence of stroke/transient ischemic attack and systemic embolism
Bleeding events; | at 2, 6, and 12 months post-procedure
  Occurrence of bleeding events
All-cause death; | at 2, 6, and 12 months post-procedure
  Occurrence of all-cause death
Cardiac death; | at 2, 6, and 12 months post-procedure
  Occurrence of cardiac death
Device-related thrombosis events; | at 2, 6, and 12 months post-procedure
  Occurrence of device-related thrombosis events
Immediate procedure success rate | Perioperation
  The occurrence rate of successful device implantation under predetermined guidance
The duration of the procedure | Perioperation
  The duration of the LAAC procedure (minutes)
the amount of contrast medium | Perioperation
  the amount of intraoperative contrast medium (ml)
the amount of radiation | Perioperation
  the amount of intraoperative radiation (Gy)
hospitalization time | Perioperation
  hospitalization time (days)
The number of replacements of the device. | Perioperation
  The number of replacements of the device.
All procedure-related complications | at 2, 6, and 12 months post-procedure
  Occurrence of all procedure-related complications
Effective LAA closure | at 2, 6, and 12 months post-procedure
  The occurrence rate of effective LAA closure (residual leak ≤5mm)

CONTACTS AND LOCATIONS:
Overall Officials: DAXIN ZHOU, MD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital,Fudan Univerisity, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No